CLINICAL TRIAL: NCT01690195
Title: Long-Term Safety and Tolerability of ABT-126 in Adults With Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors: An Open-Label Extension Study for Subjects Completing Study M11-793
Brief Title: Safety and Tolerability Study Evaluating a New Treatment for Subjects With Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data obtained from the M11-428 study is not critical to the continued evaluation of ABT-126.
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-428; 2012-000537-39 (EudraCT Number)
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ABT-126

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-126 (Experimental): ABT-126 Open-label dose
  Interventions: Drug: ABT-126

INTERVENTIONS:
Drug: ABT-126 — See arm description

SUMMARY:
This is a long term extension study to evaluate safety and tolerability of subjects who complete study M11-793 which is evaluating a new treatment for subjects with mild to moderate Alzheimer's disease on stable doses of acetylcholinesterase inhibitors.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter, 28 week extension study to evaluate the long-term safety and tolerability of ABT-126 in subjects who complete dosing through Week 24 of Study M11-793. Up to 420 subjects may participate at approximately 40 sites in seven countries.

ELIGIBILITY:
Inclusion Criteria:

* The subject and caregiver must voluntarily sign and date an informed consent. If the subject does not have the capacity to provide informed consent, full informed consent must be obtained from the subject's representative and assent must be obtained from the subject.
* The subject was randomized into Study M11-793 and completed dosing through Week 24 in that study.
* With the exception of a diagnosis of mild to moderate AD and the presence of stable medical conditions, the subject is in general good health, based upon the results of medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG.
* If male, the subject is surgically sterile (vasectomy, is sexually inactive, or is using a barrier method of birth control (condom) with spermicidal foam/gel/film/cream/suppository for the duration of the study and for 30 days following the last dose of study drug. However, if the male subject's partner has been postmenopausal for at least two years or is surgically sterile, then use of a barrier method of birth control is not required.
* The subject has an identified, reliable caregiver who will provide support and ensure compliance with the study medication and procedures, and provide accurate information about the subject's status during the study.
* The subject and caregiver must have sufficient visual, hearing and graphomotor skills to complete the study procedures.

Exclusion Criteria:

* The subject experienced an adverse event or abnormal finding in physical examination, vital signs, laboratory profile and/or ECG measurements in Study M11-793 that indicates the subject could become medically unstable during the current study.
* The subject is currently taking or is expected to be prescribed any excluded medications without the approval of Abbott medical monitor.
* The subject was noncompliant with donepezil or rivastigmine during Study M11-793 or is expected to discontinue these medications prior to conclusion of this study.
* The subject anticipates a move outside the geographic area of the investigative site or is planning extended travel inconsistent with the recommended visit intervals.
* The subject is currently enrolled in, or plans to participate in, another experimental study during the course of this trial.
* The subject developed any significant medical or psychiatric condition that, in the opinion of the investigator, renders the subject an unsuitable candidate to participate in this study.
* For any other reason the investigator considers the subject to be an unsuitable candidate to receive ABT-126 or to participate in this study.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Assessments up through 28 weeks
  Monitor each subject for clinical and laboratory evidence of adverse events on a routine basis throughout the study
Laboratory Data | Assessments up through 28 weeks
  Assessments include hematology, clinical chemistry, urinalysis and urine drug/alcohol screens
Vital Signs | Assessments up through 28 weeks
  Assessments include pulse, blood pressure and oral body temperature
Physical examinations | Assessments up through 28 weeks
  An examination of bodily functions and physical condition
Brief Neurological examination | Assessments up through 28 weeks
  Assessments include cranial nerves, motor and sensory system, reflexes, coordination, gait and station
Brief Psychiatric assessments | Assessments up through 28 weeks
  Assessments include mood, anxiety, psychosis or delusions, agitation, homicidal thoughts or behaviors
Columbia-Suicide Severity Rating Scale | Assessments up through 28 weeks
  The scale is designed to assess suicidal behavior and ideation
Cornell Scale for Depression in Dementia | Assessments up through 28 weeks
  Assesses the signs and symptoms of major depression in patients with dementia
Electrocardiogram | Assessments up through 28 weeks
  Measurements include heart rate, RR interval, PR interval, QRS duration and QT intervals

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD, Study Director — AbbVie
Locations (39):
- United States (9):
  - Site Reference ID/Investigator# 84185, Long Beach, California
  - Site Reference ID/Investigator# 84183, San Francisco, California
  - Site Reference ID/Investigator# 84187, Hamden, Connecticut
  - Site Reference ID/Investigator# 84178, Delray Beach, Florida
  - Site Reference ID/Investigator# 84180, Orlando, Florida
  - Site Reference ID/Investigator# 84186, West Palm Beach, Florida
  - Site Reference ID/Investigator# 84182, Elk Grove Village, Illinois
  - Site Reference ID/Investigator# 84181, Staten Island, New York
  - Site Reference ID/Investigator# 84179, Bennington, Vermont
- Canada (5):
  - Site Reference ID/Investigator# 84173, Gatineau
  - Site Reference ID/Investigator# 84174, Montreal
  - Site Reference ID/Investigator# 84177, Peterborough
  - Site Reference ID/Investigator# 84175, Toronto
  - Site Reference ID/Investigator# 84176, Verdun
- France (5):
  - Site Reference ID/Investigator# 84376, Dijon
  - Site Reference ID/Investigator# 84373, Limoges
  - Site Reference ID/Investigator# 84377, Paris
  - Site Reference ID/Investigator# 84374, Paris
  - Site Reference ID/Investigator# 84375, Toulouse
- Germany (6):
  - Site Reference ID/Investigator# 84382, Berlin
  - Site Reference ID/Investigator# 84380, Freiburg im Breisgau
  - Site Reference ID/Investigator# 84383, Hüttenberg
  - Site Reference ID/Investigator# 84379, Mittweida
  - Site Reference ID/Investigator# 84381, Munich
  - Site Reference ID/Investigator# 84378, Schwerin
- Greece (5):
  - Site Reference ID/Investigator# 84385, Athens
  - Site Reference ID/Investigator# 84388, Athens
  - Site Reference ID/Investigator# 84389, Athens
  - Site Reference ID/Investigator# 84386, Haidari, Athens
  - Site Reference ID/Investigator# 84390, Thessaloniki
- South Africa (5):
  - Site Reference ID/Investigator# 84395, Belville
  - Site Reference ID/Investigator# 84391, Cape Town
  - Site Reference ID/Investigator# 84393, George
  - Site Reference ID/Investigator# 84394, Johannesburg
  - Site Reference ID/Investigator# 84392, Rosebank
- United Kingdom (4):
  - Site Reference ID/Investigator# 84398, Bath
  - Site Reference ID/Investigator# 84397, Glasgow
  - Site Reference ID/Investigator# 84400, London
  - Site Reference ID/Investigator# 84399, Manchester

REFERENCES:
- [Result] Florian H, Meier A, Gauthier S, Lipschitz S, Lin Y, Tang Q, Othman AA, Robieson WZ, Gault LM. Efficacy and Safety of ABT-126 in Subjects with Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors: A Randomized, Double-Blind, Placebo-Controlled Study. J Alzheimers Dis. 2016;51(4):1237-47. doi: 10.3233/JAD-150978. PMID 26967214